CLINICAL TRIAL: NCT01859455
Title: A Randomized, Double-blind, Placebo-controlled, Single Dose, Parallel Group Study to Assess the Safety, Tolerability, Bioavailability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous LGT209 in Hypercholesterolemic Patients on Stable Doses of Atorvastatin or Simvastatin and in Healthy Volunteers
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of LGT209 in Healthy Volunteers With Elevated Cholesterol and in Hypercholesterolemic Patients Treated With Statins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLGT209X2105
Record Dates: First submitted 2013-05-09; First posted 2013-05-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-03

CONDITIONS: Hypercholesterolemia; LDL Cholesterol
Keywords: Hypercholesterolemia,; LDL cholesterol lowering,; proprotein convertase subtilisin/kexin type 9 (PCSK9),; LGT209,; drug safety,; pharmacokinetics,; pharmacodynamics
MeSH Terms: conditions — Hypercholesterolemia; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Patient: LGT209 50 mg (Experimental): 50 mg LGT209 subcutaneous (SC) (1 mL injection x 1 site) in statin patients
  Interventions: Drug: LGT209 50 mg; Drug: Statins (atorvastatin or simvastatin)
- Patient: LGT209 300 mg (Experimental): 300 mg LGT209 subcutaneous (SC) (1 mL injection x 2 sites) in statin patients
  Interventions: Drug: LGT209 300 mg; Drug: Statins (atorvastatin or simvastatin)
- Healthy Volunteers: LGT209 300 mg (Experimental): 300 mg LGT209 or placebo subcutaneous (SC) (1 mL injection x 2 sites) in healthy volunteers
  Interventions: Drug: LGT209 300 mg
- Patient: Placebo (Placebo Comparator): matching placebo subcutaneous (SC) of LGT209 50 mg or 300 mg in statin patients
  Interventions: Drug: Placebo; Drug: Statins (atorvastatin or simvastatin)
- Healthy volunteers: Placebo (Placebo Comparator): matching placebo subcutaneous (SC) of LGT209 300 mg in healthy volunteers
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LGT209 50 mg — Active experimental drug
  Arms: Patient: LGT209 50 mg
Drug: LGT209 300 mg — Active experimental drug
  Arms: Healthy Volunteers: LGT209 300 mg; Patient: LGT209 300 mg
Drug: Placebo — Placebo comparator
  Arms: Healthy volunteers: Placebo; Patient: Placebo
Drug: Statins (atorvastatin or simvastatin) — Stable doses of atorvastatin or simvastatin
  Other Names: Atorvastatin; Simvastatin
  Arms: Patient: LGT209 300 mg; Patient: LGT209 50 mg; Patient: Placebo

SUMMARY:
This study is designed to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of LGT209 in hypercholesterolemic patients taking common statin medications and in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Male and female subjects 18 to 70 years of age, in general good health with fasting LDL-cholesterol >90 mg/dL and fasting serum triglycerides <400 mg/dL
* Patients on statin therapy: Male and female patients 18 to 70 years of age receiving atorvastatin or simvastatin and with fasting LDL-cholesterol >90 mg/dL and fasting serum triglycerides <400 mg/dL

Exclusion Criteria:

Healthy volunteers:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Women of child-bearing potential unless using highly effective methods of contraception
* Conditions which might impact the safety or biologic activity of the study drug

Statin patients:

* Use of concomitant medications known to impact the safe use or efficacy of atorvastatin and simvastatin based on drug labels
* Women of childbearing potential unless using highly effective methods of contraception during dosing and for at least 100 days after study drug administration
* Conditions which might impact the safety or biologic activity of the study drug

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects (patients and healthy volunteers) with adverse events, serious adverse events and death | 12 weeks
Plasma concentrations of LGT209 following subcutaneous administration | 12 weeks
Change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) concentration | baseline and 12 weeks
Change from baseline in low density lipoprotein-cholesterol (LDL-C) concentration | baseline and 12 weeks

SECONDARY OUTCOMES:
Plasma concentrations of atorvastatin in patients | 2 weeks
Plasma concentrations of simvastatin in patients | 2 weeks
Serum concentrations of PCSK9 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Miramar, Florida

REFERENCES:
- See also: Results for CLGT209X2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8686